CLINICAL TRIAL: NCT00754936
Title: ERPs, Cognitive Dysfunction and Treatment Response of Geriatric Depression
Brief Title: Treatment Response of Geriatric Depression
Acronym: ERP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0703009061; R01MH079414-01A1 (NIH)
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-02

CONDITIONS: Depression
Keywords: Depression
MeSH Terms: conditions — Depression | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Escitalopram (Experimental): 12 week open label with 2 week placebo period (14 weeks total)
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — 20 mg by mouth daily
  Other Names: Lexapro

SUMMARY:
The purpose of this study is to examine the relationship between brain electrical activity in elderly depressed patients and response to antidepressant medication treatment. Elderly patients with depression will be treated for 12 weeks with an antidepressant medication commonly used in clinical practice called escitalopram (Lexapro). Brain electrical activity will be assessed using electrophysiological tests. Researchers are interested in whether the brain electrical activity of elderly people with depression before they start the medication can tell us who amongst them will improve with antidepressant treatment and to what extent. They will also determine whether patients' brain electrical activity during the 12 weeks of medication treatment will change in any way and whether this change will be linked with a change in the severity of their depression. Researchers hope that information gained from this study will help to better understand the brain processes associated with depression and its successful treatment.

DETAILED DESCRIPTION:
This research study will examine how the brain electrical activity of elderly depressed patients is related to how quickly and how well they respond to antidepressant medication treatment. Brain electrical activity will be assessed using electrophysiological tests. Elderly patients with depression will be treated for 12 weeks with an antidepressant medication commonly used in clinical practice called escitalopram (Lexapro). Before they start treatment, patients will be asked questions about their depression to measure how severe it is. They will also be asked to have their brain electrical activity recorded while they perform tests on a computer screen. The questions about their depression and the brain electrical recordings will be repeated regularly during the 12 weeks they will be treated with antidepressant medication. The researchers are interested to see whether the brain electrical activity of elderly people with depression before they start the medication can tell us who amongst them and to what extent will finally improve with treatment with escitalopram (Lexapro). They will also determine whether patients' brain electrical activity, during the 12 weeks they will be receiving the medication treatment, will change in any way and whether this change will be linked with the change in the severity of their depression. It is hoped that information gained from this study will help the investigators to better understand the brain processes associated with depression and its successful treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Major depression, unipolar without psychotic features (by DSM-IV criteria) -Severity of depression: A 24-Item HDRS above 19 at screening and at baseline -
* Level of Executive Dysfunction: Two strata within each age stratum: Stroop Color-Word scores - one half of the sample < 26, one of half ≥ 26.
* Capacity to provide informed consent.

Exclusion Criteria:

* High suicide risk, i.e. intent or plan to attempt suicide in near future
* Presence of any current Axis I psychiatric disorder (other than unipolar major depression or specific phobias) including substance abuse (those with a history of substance abuse must be abstinent for at least 3 months prior to entry)
* Axis II diagnosis of antisocial personality disorder, mental retardation and pervasive developmental disorder (DSM-IV)
* History of psychiatric disorders such as psychotic depression, primary psychotic disorder, or bipolar spectrum disorder (bipolar disorder and hypomania are exclusions)
* Cognition: MMSE scores below 24 or diagnosis of dementia by DSM-IV
* Acute or severe medical illness, i.e., delirium, metastatic cancer, decompensated cardiac, liver or kidney failure, major surgery, stroke or myocardial infarction during the three months prior to entry; or drugs known to cause depression, e.g., reserpine, alpha-methyl-dopa, steroids, sympathomimetics withdrawal
* Presence of a significant neurological disease such as Parkinson's disease, primary or secondary seizure disorders, intracranial tumors, severe head trauma; neurodegenerative diseases i.e. MS
* History of failure to respond to escitalopram (Lexapro) (20mg/day for 6 weeks or longer) during the current or previous depressive episodes
* History of intolerance to escitalopram (Lexapro) or use of concomitant drugs that may provide reason to believe that escitalopram is contraindicated. Active treatment with fluoxetine at the time of screening
* Patients' unwillingness or inability to gradually withdraw all other psychotropic medications (except for the following: Low and stable doses of opiates and non-benzodiazepine hypnotics (e.g. zolpidem (5 or 10 mg), zaleplon (5 or 10 mg), or eszopiclone (1 or 2 mg).Low and stable doses of diazepam and other anxiolytics should be tapered at screening; inability to tolerate taper is not an exclusion criteria.
* Inability to perform any of the ADLs (MAI: ADL subscale) even with assistance, e.g. walking with a cane is not an exclusion criterion
* Inability to speak English
* Aphasia

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Alexopoulos, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College-Westchester Division, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall flow of study participants
Pre-assignment Details: 106 participants enrolled in the study; however, 35 exited during the 2-week washout period and did not start study medication.
Period: Overall Study
Arm/Group | Escitalopram
Started | 71
Completed | 59
Not Completed | 12
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2
Not completed — Side Effects | 3
Not completed — Inter-current medical events | 3

BASELINE CHARACTERISTICS:
Arm/Group | Escitalopram
Number analyzed (Participants) | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.91 (7.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 67
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 66
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 71
Hamilton Depression Rating Scale (HDRS) 24-Item Total Score [Mean (Standard Deviation); unit: units on a scale] — HDRS 24 item: scores can range from 0-76; higher is worse(more depressed)
  units on a scale | 23.83 (4.48)
Montgomery and Asberg Depression Rating Scale (MADRS) Total Score [Mean (Standard Deviation); unit: units on a scale] — MADRS: scores can range from 0-60; higher is worse(more depressed)
  units on a scale | 24.08 (5.74)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Rating Scale (Depression Severity)
Description: A published and widely used scale for measuring severity of depression. Montgomery Asberg Depression Rating Scale scores can range from 0-60. Higher scores indicate greater severity of depression. Total scores are reported with no subscales.
Time Frame: 14 weeks from enrollment (12 weeks from medication start)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram
Number analyzed (Participants) | 71
units on a scale | 12.23 (7.67)

2. Secondary Outcome: Hamilton Depression Rating Scale (Depression Severity)
Description: A published and widely-used scale for rating depression severity, the Hamilton Depression Rating Scale 24 item total scores range from 0-76. Higher scores indicate greater severity of depression. Total scores are reported with no subscales.
Time Frame: 14 weeks from enrollment (12 weeks from medication start)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram
Number analyzed (Participants) | 71
units on a scale | 11.47 (6.64)

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | Escitalopram
All-Cause Mortality (participants affected / at risk) | 0/71
Serious Adverse Events (participants affected / at risk) | 3/71
Other Adverse Events (participants affected / at risk) | 47/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram (N=71)
Hospitalisation (Surgical and medical procedures) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram (N=71)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Burning sensation (Nervous system disorders) | 2 (3)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
Colonoscopy (Investigations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 12 (15)
Dizziness (Nervous system disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 21 (38)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Groin infection (Infections and infestations) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Sinus headache (Nervous system disorders) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Surgery (Surgical and medical procedures) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes